CLINICAL TRIAL: NCT07393087
Title: Jafron Cytokine Adsorber During Pediatric Open-Heart Surgeries
Acronym: JACKPOT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Antoine Schneider, Principal Investigator, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CER-VD-2025-D0097
Record Dates: First submitted 2026-01-22; First posted 2026-02-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Surgery Recovery; Inflammation; Complex Cardiovascular Surgery With Cardiopulmonary Bypass; Cytokine Storm; Pediatric Open Heart Surgery
Keywords: Feasibility pilot study; Pediatric open heart surgery; Hemoadsorption
MeSH Terms: conditions — Inflammation; Cytokine Release Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemoadsorption (Experimental): Cardiopulmonary bypass (CPB) will be conducted as per institutional protocols and an HA-60® cartridge (Jafron Biomedical, Guangdong, China) will be inserted within the circuit for hemoadsorption.
  Interventions: Device: Hemoadsorption
- Control (No Intervention): Cardiopulmonary bypass will be conducted as per institutional protocols, without hemoadsorption (standard-of-care)

INTERVENTIONS:
Device: Hemoadsorption — The hemoadsorption treatment will be performed during the entire duration of the CPB. The blood flow within the hemoadsorber will be controlled and set to 7% of the theoretical minimal CPB flow which is calculated as 2.5 L/min/1.73m2 of body surface area.
  Arms: Hemoadsorption

SUMMARY:
This prospective single-center randomized controlled trial aims at evaluating the safety and feasibility of an hemoadsorption protocol using Jafron HA-60 during cardio-pulmonary bypass in 20 pediatric patients undergoing open-heart surgery.

DETAILED DESCRIPTION:
Cardiopulmonary bypass (CPB) is an extracorporeal system that temporarily takes over the functions of the heart and lungs by diverting blood during cardiac surgery. However, the use of CPB is know to trigger a significant systemic inflammatory response, largely mediated by cytokines. In severe cases, this response may result in vasoplegia, hypotension, and subsequent organ dysfunction. Several pharmacological interventions have been investigated to reduce the incidence and severity of this post-surgical inflammatory response, but results have been very mitagated. Among emerging strategies, the pre-procedural removal of circulating cytokines through hemoadsorption represents a promising approach. In particular the use of a HA-60® cartridge (Jafron Biomedical, Guangdong, China) integrated into the CPB circuit may help attenuate the inflammatory cascade.

This pilot study is designed to evaluate the feasibility and safety of implementing an hemoadsorption protocol during cardiopulmonary bypass in a pediatric population. Pediatric patients scheduled for complex cardiac procedures will be enrolled before surgery and randomly assigned in a 1:1 ratio to either receive hemoadsorption therapy with standard care (intervention group) or standard care alone (control group).

In the intervention group, an HA-60® hemoadsorption cartridge will be integrated into the CPB circuit during setup and used throughout the duration of the bypass. Four blood samples will be collected : Post-anestesia induction, CPB termination, ICU admission, and 24 hours post ICU admission-to measure cytokine levels. Clinical data, including vital signs, organ support, demographics, and medical history, will be recorded in the electronic medical records.

ELIGIBILITY:
Inclusion Criteria:

* Children ≤ 10 years old at study inclusion
* Children weighing at least 5 kg at study inclusion
* Planned for open-heart cardiac surgery with CPB-time ≥ 120 min and aortic clamping.
* Informed consent obtained from parent(s)/legal representative

Exclusion Criteria:

* Children having an indication to receive hemoadsorption during CPB for drugs removal or other medically justified reason
* Previous enrolment into the current study
* Off-pump procedure
* Chronic immunosuppression (chronic corticosteroid therapy, chemotherapy, anti-leucocyte drugs, TNF blockers or else)
* Known allergy to heparin or heparin induced thrombocytopenia.
* Severe thrombopenia (platelets count before surgery < 20G/L)
* Parent(s)/legal representative not able to understand/read French and/or English
* Participation in another conflicting research study

Max Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Screened-to-enrolled patients' ratio and number of intervention delivery group | Start CPB, End CPB, 1 Day and aftrer 28 day
  * Screened-to-enrolled patients' ratio ≥ 0.3*
  * ≥ 80% of intervention delivery in intervention group (number of patients who received hemoadsorption > 50% of CPB duration)
  * Duration of recruitment: no more than 36 months (approximately 0.56 patient per month)
  * <5% of study interruptions attribuable to insufficiant resources or logistical constraints *(Previous pilot studies in intervention contexts report screened-to-enrolled patient ratios of approximately 0.30-0.50; therefore a threshold of ≥ 0.30 has been chosen as a minimal acceptable benchmark for feasibility.)
Device-related adverse events | From beginning of cardiopulmonary bypass to 7 days after ICU admission or ICU discharge wichever occurs first.
  Assessed with the occurrence of 4 categories of adverse events in each group:
  Device-related complications:
  • Technical failure to perform the treatment: thrombosis of the cartridge, circuit leak or inability to perform the treatment for all CPB duration.
  Tolerance:
  * New allergic or anaphylactoid reaction (stage ≥ 2 by H. L. Mueller [5])
  * New fever (> 39°C for more than an hour).
  Bleeding/haematological complications*:
  * Intracranial haemorrhages
  * Need for massive transfusion (>10mL/kg/h during more than 3 consecutive hours)
  * Incidence of new thrombocytopenia (mild <150 G/L, moderate, <100 G/L severe < 50 G/L) *(We will consider separately bleeding/haematological complications occurring during the procedure (from CPB initiation to ICU admission) and those occurring from ICU admission to day 7 or ICU discharge, whichever occurs first.)
  All other event judged relevant by the investigator (i.e. cardiac arrest). NB: "New" means not present at the time of CPB initiation

SECONDARY OUTCOMES:
Pediatric Logistic Organ Dysfunction-2 (PELOD-2) score at 24 hours | Measured between post-anestesia induction and 24 hours post ICU-admission
  Difference in the PELOD-2 score between before surgery and 24 hours after admission to intensive care. The PELOD-2 score ranges from a minimum of 0 (indicating no organ dysfunction) to a maximum of 33 (indicating the most severe level of organ dysfunction)
Pediatric Logistic Organ Dysfunction-2 (PELOD-2) worst value | Within 4 hours of ICU admission
  Efficacy measured by the PELOD-2 worst value between admission to intensive care and 24 hours after admission to intensive care. The PELOD-2 score ranges from a minimum of 0 (indicating no organ dysfunction) to a maximum of 33 (indicating the most severe level of organ dysfunction)
Pediatric Logistic Organ Dysfunction-2 (PELOD-2) score at 48 hours | Measured between 24 hours and 48 hours after ICU admission
  PELOD-2 difference between groups in the PELOD-2 score measured between 24 hours and 48 hours after ICU admission. The higher the PELOD-2 the highest the probability of death.The PELOD-2 score ranges from a minimum of 0 (indicating no organ dysfunction) to a maximum of 33 (indicating the most severe level of organ dysfunction).
Change in cytokine levels compared to baseline | at the end of CPB, at the admission in ICU and 24 hours after ICU admission
  Relative and absolute change in the plasma levels of cytokines at different timepoints, compared with their levels at baseline (post-anestesia induction).
ICU and hospital lenght of stay | At time of hospital discharge, an average 20 days after ICU admission
  Lengths of stays, in days
ICU, hospital, and 28 days (from ICU admission) mortality | At time of hospital discharge, an average 20 days after ICU admission and up to 28 days after ICU admission
  All-cause mortality
Days alive without respiratory support | At day 28 from ICU admission
  Number of days alive and without mechanical ventilation
Days alive without renal replacement therapy | At day 28 from ICU admission]
  Number of days alive and without renal replacement therapy
Days alive without vasopressors | At day 28 from ICU admission]
  Number of days alive and without vasopressors
Days alive without ECMO support | At day 28 from ICU admission
  Number of days alive and without Extracorporeal membrane oxygenation (ECMO)
Post-operative complications | At time of ICU discharge, up to 7 days after ICU admission
  Post-operative Acute Kidney Injury, transfusion of red blood cells, sepsis, liver injury

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Schneider, MD-PhD, Principal Investigator — Centre Hospitalier Universitaire Vaudois (CHUV) and University of Lausanne
Locations (1):
- Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No